CLINICAL TRIAL: NCT02929433
Title: Conservative Treatment of Rotator Cuff Tear: The Role of Cycloergometer
Brief Title: Cycloergometer and Rotator Cuff Tear
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fondazione Salvatore Maugeri (Other)
Responsible Party: Principal Investigator, Bernardo Gialanella, Doctor, Fondazione Salvatore Maugeri
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: cts 2012-13
Record Dates: First submitted 2016-09-28; First posted 2016-10-11 (Estimated); Last update posted 2016-10-11 (Estimated); Status verified 2016-10

CONDITIONS: Rotator Cuff Tear
Keywords: disability; pain; Rotator Cuff Tear; rehabilitation; range of motion (ROM)
MeSH Terms: conditions — Rotator Cuff Injuries; Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Cycloergometer group (Experimental): Training at home with the cycloergometer per 20 minutes twice a day. The protocol suggested a continous use of the cycloergometer for a period of 6 months after 2 weeks of rehabilitation as outpatient.
  Interventions: Other: Cycloergometer
- Control group (No Intervention): Usual care after a period (2 weeks) of rehabilitation as outpatient.

INTERVENTIONS:
Other: Cycloergometer — Daily training of the RCT patients was provided by the use of a cycloergometer at home. Educational support once a month was guaranteed by a nurse of the telemedicine service
  Arms: Cycloergometer group

SUMMARY:
The cycloergometer is a mechanical device consisting of a bicycle frame fixed on a support base, designed to measure the amount of muscle work performed during exercise and the resistance to pedaling. The cycloergometer has been already employed in many fields of medicine.

However, up to date, a little use of cycloergometer in the management of chronic joint diseases has been documented and scientific studies have not clarified if cycloergometer is effective in these diseases and, particularly, in Rotator Cuff Tear patients.

DETAILED DESCRIPTION:
To evaluate the effects of cycloergometer on pain during activities (primary outcome) and shoulder functionality, the investigators performed a prospective randomized controlled study (pilot study) in patients with a symptomatic full-thickness RCT.

Since cycloergometer works through a continuous active and passive joint mobilization, the investigators expect it can reduce pain and improve shoulder functionality becoming a useful tool for physicians in the management of RCT patients.

ELIGIBILITY:
Inclusion Criteria:

* positive imaging diagnosis of full-thickness RCT
* surgery not considered as the first treatment of choice
* willingness to sign the informed consent form.

Exclusion Criteria:

* inflammatory rheumatic diseases
* history of fracture or operations around the shoulder region
* neurological diseases
* infections or tumours
* diabetes
* coagulation diseases
* intra-articular injections of the involved shoulder within the last 12 months.

Min Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 38 (Actual)
Dates: Start 2013-01; Primary Completion 2014-12 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
Visual Numeric Scale (VNS) | Change from Baseline VNS at 6 months after the out-patient rehabilitation
  The scale evaluated shoulder pain during activity

SECONDARY OUTCOMES:
Constant-Murley scale | Change from Baseline Constant-Murley scale at 6 months after the out-patient rehabilitation
  The scale evaluated shoulder functionality
Health Assessment Questionnaire (HAQ) | Change from Baseline HAQ at 6 months after the out-patient rehabilitation
  The Questionnaire evaluated Disability

CONTACTS AND LOCATIONS:
Overall Officials: Bernardo Gialanella, MD, Principal Investigator — Fondazione Salvatore Maugeri

IPD SHARING:
Plan to Share IPD: Yes
Scientific manuscript